CLINICAL TRIAL: NCT05292456
Title: Monıtorıng Glucocortıcoıd Treatment Using Glucocorticoid Toxicity Index (GTI) In Patıents Followed In Rheumatology Clınıc
Brief Title: Monıtorıng Glucocortıcoıd Treatment In Patıents Followed In Rheumatology Clınıc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Melda Bahap, Principal investigator, Hacettepe University
Other Study IDs: KA- 21026
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Glucocorticoids Toxicity; Rheumatoid Arthritis; Vasculitis; Systemic Lupus Erythematosus
Keywords: glucocorticoid toxicity index; Drug-Related Problem; Glucocorticoid; Rheumatoid Arthritis; Vasculitis; Clinical Pharmacist
MeSH Terms: conditions — Arthritis, Rheumatoid; Vasculitis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA, SLE, and vasculitis patients who have just started glucocorticoid treatment
- RA, SLE and vasculitis patients receiving glucocorticoid treatment for the last 2 years

SUMMARY:
Hypothesis 1: A reduction in side effects is achieved with monitoring glucocorticoid treatment by using the Glucocorticoid Toxicity Index (GTI) in patients using glucocorticoids.

Hypothesis 2: Monitoring treatment by using GTI in patients using glucocorticoids causes a decrease in glucocorticoid toxicity and an increase in the quality of life of patients.

Hypothesis 3: With the involvement of the clinical pharmacist in the multidisciplinary team in patients using glucocorticoids, the drug-related problems of the patients are detected and prevented.

The aim of this study was to evaluate the glucocorticoid treatment of patients with RA, SLE and vasculitis treated with glucocorticoids prospectively by a multidisciplinary team with GTI. In addition, it was aimed to identify and prevent drug-related problems by reviewing all drugs used in these patients by the clinical pharmacist.

DETAILED DESCRIPTION:
In this study, the side effects of glucocorticoids used by patients will be evaluated using the Glucocorticoid Toxicity Index (GTI) index. This index includes areas for commonly recognized adverse events as a result of cumulative steroid exposure. It is weighted and measures both worsening and improvement. Scores range from -346 to 439 with cumulative worsening score relating to an increase in GC toxicity burden. "-" points indicate improvement, "+" points indicate worsening. The higher the patient's burden of glucocorticoid toxicity, the higher his score.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Individuals who have received glucocorticoid treatment for RA, SLE or vasculitis in the last 2 years or at current admission.
* Patients approved by the physician to participate in the study
* Patients giving written consent

Exclusion Criteria:

* Younger than 18
* Patients with communication disabilities
* Patients involved in another clinical and/or drug trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of RA, SLE or vasculitis followed in the Hacettepe University Hospitals Rheumatology Outpatient Clinic and receiving glucocortioid therapy will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
change in Glucocorticoid Toxicity Index (GTI) scores | Each patient will be followed up for a total of 6 months, at 3 and 6 months.
  In this study, it is predicted that a change in GTI scores will be achieved during 3-month follow-up in patients with long-term and newly diagnosed RA, SLE and vasculitis. When the 6-month follow-up of each patient is completed, the study will be terminated.
  In this study, the side effects of glucocorticoids used by patients will be evaluated using the Glucocorticoid Toxicity Index (GTI) index. This index includes areas for commonly recognized adverse events as a result of cumulative steroid exposure. It is weighted and measures both worsening and improvement. Scores range from -346 to 439 with cumulative worsening score relating to an increase in GC toxicity burden. "-" points indicate improvement, "+" points indicate worsening. The higher the patient's burden of glucocorticoid toxicity, the higher his score.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Karadag, prof. doctor, Study Director — Hacettepe University Faculty of Medicine, Department of Internal Medicine, Division of Rheumatology,
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)